CLINICAL TRIAL: NCT05544968
Title: A Phase I Study to Investigate the Safety, Tolerability, and Preliminary Efficacy of Anti-CD30 Bispecific Antibody-Armed Anti-CD3-Activated Autologous T-Cells (CD30 biAb-AATC) in Patients With Relapsed/Refractory CD30 Positive Hematopoietic Malignancies
Brief Title: Anti-CD30 biAb-AATC in Patients With Relapsed/Refractory CD30 Positive Hematopoietic Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Guru Subramanian Guru Murthy, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00052928
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hodgkin Disease; CD30-Positive Diffuse Large B-Cell Lymphoma; CD30+ Anaplastic Large Cell Lymphoma; CD30+ Pleomorphic Large T-Cell Cutaneous Lymphoma; CD30+ Immunoblastic Large T-Cell Cutaneous Lymphoma; Leukemia; Lymphoma
Keywords: CD30; Cancer; Bispecific; Cellular Therapy; T Cell; autologous; relapse; refractory
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Leukemia; Lymphoma; Neoplasms; Recurrence | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- CD30biAb-AATC (Dose Level -1 -- 40 x 10^6 cells/kg/infusion + GM-CSF 250 μg/m^2) (Experimental): Patients will undergo weekly administration of dose escalating CD30 biAb-AATC infusions with twice weekly subcutaneous GM-CSF (250 μg/m^2) in 4-week cycles for a maximum of two total cycles.
  A standard 3+3 dose escalation design will be utilized for this study.
  Interventions: Drug: anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells (CD30 biAb-AATC); Drug: GM-CSF
- CD30biAb-AATC (Dose Level 1 -- 80 x 10^6 cells/kg/infusion + GM-CSF 250 μg/m^2) (Experimental): Patients will undergo weekly administration of dose escalating CD30 biAb-AATC infusions with twice weekly subcutaneous GM-CSF (250 μg/m^2) in 4-week cycles for a maximum of two total cycles.
  A standard 3+3 dose escalation design will be utilized for this study.
  Interventions: Drug: anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells (CD30 biAb-AATC); Drug: GM-CSF
- CD30biAb-AATC (Dose Level 2 -- 120 x 10^6 cells/kg/infusion + GM-CSF 250 μg/m^2) (Experimental): Patients will undergo weekly administration of dose escalating CD30 biAb-AATC infusions with twice weekly subcutaneous GM-CSF (250 μg/m^2) in 4-week cycles for a maximum of two total cycles.
  A standard 3+3 dose escalation design will be utilized for this study.
  Interventions: Drug: anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells (CD30 biAb-AATC); Drug: GM-CSF
- CD30biAb-AATC (Dose Level 3 -- 160 x 10^6 cells/kg/infusion + GM-CSF 250 μg/m^2) (Experimental): Patients will undergo weekly administration of dose escalating CD30 biAb-AATC infusions with twice weekly subcutaneous GM-CSF (250 μg/m^2) in 4-week cycles for a maximum of two total cycles.
  A standard 3+3 dose escalation design will be utilized for this study.
  Interventions: Drug: anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells (CD30 biAb-AATC); Drug: GM-CSF
- CD30biAb-AATC Recommended Phase 2 Dose (RP2D) (Experimental): The RP2D is defined as the dose level below the dose where two or more dose-limiting toxicities were observed.
  Interventions: Drug: anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells (CD30 biAb-AATC); Drug: GM-CSF

INTERVENTIONS:
Drug: anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells (CD30 biAb-AATC) — anti-CD30 Bispecific Antibody-armed anti-CD3-Activated Autologous T-cells
  Other Names: CD30 biAb-AATC
Drug: GM-CSF — Hematopoietic agent that helps form white blood cells.
  Other Names: granulocyte-macrophage colony-stimulating factor; sargramostim

SUMMARY:
This first-in-human trial will assess the safety, feasibility, and efficacy of an immunotherapy with a novel CD30 antibody conjugated to a CD3 antibody that is preloaded onto a patient's own T-cells, generating a CD30 bispecific antibody-armed, anti-CD3-activated, autologous T-cells (CD30 biAb-AATC).

DETAILED DESCRIPTION:
Non-randomized, single arm, dose escalating, Phase I study evaluating the feasibility and safety of a novel anti-CD30 biAb-AATC product for adult patients with relapsed/refractory CD30+ cancer. Following T-cell collection patients are recommended to receive a bridging chemotherapy for 21 days while product is being generated and quality control assessed. Patients will then undergo weekly administration of dose escalating CD30 biAb-AATC infusions with twice weekly subcutaneous GM-CSF in 4-week cycles for a maximum of two total cycles.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: Patients must have had histologic or cytologic verification of the below qualified malignancy. The pathology report for the diagnosis under which the patient is being enrolled and associated molecular diagnostic reports must be submitted.

a. Hodgkin's Lymphoma (HD): Patients with HD are eligible with one of the following:

i. Second or greater recurrence or refractory to at least 2 prior therapeutic regimens.

ii. Any relapse after HSCT.

b. Non-Hodgkin Lymphoma (NHL): Patients with NHL are eligible with one of the following:

i. Second or greater recurrence or refractory to at least 2 prior therapeutic regimens.

ii. Any relapse after HSCT or CAR T cell therapy.

c. Acute Myeloid Leukemia (AML): Patients with AML are eligible with one of the following:

i. First or greater relapse.

ii. Primary refractory disease with at least 1 prior induction attempts.

d. Acute Lymphoblastic Leukemia (ALL): Patients with ALL are eligible with one of the following:

i. Second or greater relapse or refractory to at least 2 prior therapeutic regimens.

ii. Any relapse after HSCT or CAR T cell therapy.

e. Other Hematopoietic malignancy not listed above for which standard curative measures do not exist, are not proven to prolong survival with an acceptable quality of life, or are no longer effective.

CD30 Expression Status: Disease specific histologic, cytologic, or Fluorescence-Activated Cell Sorting (FACS)-confirmed CD30 cell surface expression on malignant cells is required. CD30 surface expression must be confirmed at most recent histologic, cytologic, or FACS assessment of disease. This confirmation must occur at recurrence. No repeat CD30 expression verification is required for patients with primary refractory diseases. Pathology and diagnostic reports verifying the CD30 expression status must be submitted.

Leukemia CD30 Expression Criteria: Flow cytometry immunophenotypic analysis of bone marrow or peripheral blood. Surface expression of CD30 expression on blasts "positive" with ≥20% expression consistent with established precedents.

Lymphoma CD30 Expression Criteria: Flow cytometry immunophenotypic analysis of lymphoma sample or immunohistochemical assessment of formalin-fixed paraffin embedded sample. Flow cytometry assessment surface expression or immunohistochemical membranous expression of CD30 on neoplastic cells "positive" with ≥ 1% expression consistent with established precedents.

Disease Status:

i. Lymphomas: Patients must have measurable disease for assessment of radiographic response defined as either nodal disease >/=1.5 cm or extranodal lesion >/=1.0 cm.

ii. Leukemias: Patients must have relapsed/refractory (including MRD >0.01% by flow cytometry) disease.

Prior Therapy: Patients must have recovered from the acute toxic effects of prior anticancer chemotherapy, defined as resolution of all such toxicities to ≤ Grade 2 or lower prior to entering this study and initiating lymphocyte collection.

i. Myelosuppressive chemotherapy: Patients must not have received myelosuppressive therapy within 3 weeks of apheresis for this study.

ii. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g., Neulasta) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.

iii. Biologic (anti-neoplastic agent): At least 7 days after the last of a biologic agent that is not a monoclonal antibody and infusion of study product on this study. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.

iv. Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g., tumor vaccines or CAR T-cell therapy.

v. Monoclonal antibodies: At least 3 half-lives must have elapsed after treatment with a monoclonal antibody and infusion of study product on this study.

vi. XRT: >2 weeks must have elapsed for XRT and infusion of study product.

vii. Prior treatment with etoposide, vincristine, CD30 targeted agent, or a bispecific antibody-armed activated autologous T-cell product as single agents or in combination are eligible for this study provided there were no known hypersensitivity or allergic reactions attributed to any of the components of compounds of similar composition to etoposide, vincristine, CD30 targeted agent, or a bispecific Antibody-armed activated autologous T cell product.

Age: Patients must be ≥ 18 years at time of study enrollment.

Life Expectancy: Life expectance of >12 weeks.

Performance Status: Karnofsky ≥50% for patients. Note: Neurologic deficits in patients with CNS involvement must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Organ Function Requirements: Have acceptable organ function as defined below:

i. Renal: Serum creatinine concentration ≤1.5 × institutional upper limit of normal (ULN) based on the age and sex, or creatinine clearance (CrCl) ≥50 mL/min (as measured by Cockcroft-Gault formula or acceptable equivalent).

ii. Hepatic:

1. Direct Bilirubin <1.5 x upper limit of normal (ULN) for age. For patients with documented Gilbert's syndrome (unconjugated hyperbilirubinemia) the bilirubin must be ≤3 x ULN for age.
2. SGPT (ALT) <3 x ULN.
3. Serum albumin >2 g/dL.

iii. Pulmonary: Pulse oximetry >90% on room air. Subjects must have no supplemental oxygen requirement.

iv. Cardiac: LVEF ≥ 40% by ECHO or MUGA.

v. HL and NHL specific criteria: Bone Marrow:

Adequate bone marrow reserves as evidenced by the following: For patients with lymphoma without known bone marrow involvement:

i. Peripheral absolute neutrophil count (ANC) ≥1,000/mm^3.

ii. Platelet count ≥50,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).

b. For patients with known bone marrow disease or lymphoma with known bone marrow involvement will be eligible for study provided they meet the following transfusion criteria.

i. Eligible regardless of ANC, hemoglobin or platelet counts provided they respond to red cell or platelet transfusions.

ii. They will not be eligible for assessment of hematologic toxicity.

Pregnancy: It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below.

1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 7 days prior to enrollment.
2. Female patients must meet one of the following:

i. Postmenopausal for at least one year before the screening visit, or ii. Surgically sterile, or iii. If they are of childbearing potential, agree to practice a reliable method of contraception from the time of signing of the informed consent form through three months after the last dose of study drug. OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)

c. Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

i. Practice effective barrier contraception during the entire study treatment period and through three months after the last study drug dose, OR agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

Consent: Ability to under understand a written informed consent document, and the willingness to sign it. Voluntary written consent will be documented before initiation of study-related procedures not part of normal medical care. Consent may be withdrawn by the subject/guardian without prejudice to future medical care.

Exclusion Criteria

Prior Therapy: Any toxicities from prior treatment, >Grade 3 per CTCAE v5.0 Hematopoietic stem cell transplantation (HCT) or chimeric antigen receptor T-cell therapy (CAR-T cell) within 60 days of enrollment, or evidence of veno-occlusive disease (VOD) at any time post-transplant.

Investigational Agent: Treatment with any investigational agent within 14 days of enrollment.

Exclusion Requirements Due to Comorbid Disease or Concurrent Illness:

Immune: Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Steroid premedication for imaging scans is allowed. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

Infectious: Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment). Patients with possible fungal infections must have had appropriate anti-fungal antibiotics and adequately controlled. HIV-positive patients on combination antiretroviral therapy are ineligible because of the unknown ability to expand T cell populations for CD30 biAb-AATC product in this setting. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Pulmonary: Prior history of anti-CD30 therapy related pulmonary toxicity.

Neurologic: Prior history of progressive multifocal leukoencephalopathy (PML).

Cardiac: Patients diagnosed with NYHA Class III or IV congestive heart failure, ventricular arrhythmias, or uncontrolled hypertension.

Allergies: Known hypersensitivity or allergic reaction attributed to any of the components of CD30 biAb-AATC or to compounds of similar composition to CD30 targeted agent, or a bispecific Antibody-armed activated autologous T cell product.

Pregnant or Breastfeeding: Pregnant or breastfeeding females will not be allowed to enroll on this study. Female patients with infants must agree not to breastfeed their infants during the entire study treatment period and through three months after the last study drug dose. Agents used in this study are known to be teratogenic to a fetus. There is there is no information on the excretion of CD30 biAb-AATC agents into breast milk but potential risk for adverse events in nursing infants secondary to treatment of the mother with a CD30 biAb-AATC.

Secondary Malignancy: Patients should not have a history of any second malignancy in the last 1 year with exception of the diagnosis for inclusion; subjects with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Subjects with other malignancies are eligible if they have been continuously disease free for at least 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 years
  To determine the MTD and recommended Phase II dose of CD30 biAb-AATC administered once weekly for a total of 4 doses per cycle

CONTACTS AND LOCATIONS:
Overall Officials: Guru Subramanian Guru Murthy, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No